CLINICAL TRIAL: NCT03299673
Title: Observational Study to Investigate the Compliance of Patients With COPD With the 8-item Morisky Medication Adherence Scale and Assessing the Quality of Life of Patients as Shown by the Clinical COPD Questionnaire (CCQ) Questionnaire.
Brief Title: AdHerencE to Treatment and quAlity of Life in COPD
Acronym: AHEAD
Status: Completed | Type: Observational
Sponsor: Elpen Pharmaceutical Co. Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2017-HAL-EL-75
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Chronic Obstructive Pulmonary Disease; Compliance, Patient; Quality of Life
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Patient Compliance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The present non-interventional observational study in the Greek population aims at collecting the characteristics of COPD patients selected to be given the inhaled combination of fluticasone propionate and salmeterol in doses of 100 μg mcg (250 μg) mcg (500 g) mcg through the Elpenhaler® device, to investigate (a) the effectiveness of the treatment for compliance and the quality of life of the patients; and (b) the safety of the drugs in patients whose disease is treated either in a hospital or in a private physician.

DETAILED DESCRIPTION:
Rolenium® is an inhalable combination the active ingredients of which is the inhaled combination of fluticasone propionate and salmeterol in doses (100 + 50) mcg, (250 + 50) mcg, (500 + 50) mcg administered via the Elpenhaler ®, developed by ELPEN. It has been approved as a bronchodilator therapy for COPD (a fast-exiting volume in the first second (FEV1) after a bronchodilator less than 60% predicted) with a history of repeated seizures that have significant symptoms despite regular bronchodilator therapy. For COPD in adults an inhalation of 500 micrograms of fluticasone propionate and 50 micrograms of salmeterol twice daily is recommended4. More information on the efficacy and safety of the investigational medicinal product is provided in the Summary of Product Characteristics (SPC).

ELIGIBILITY:
Inclusion Criteria:

* Patients to be started on Rolenium®, an inhaled combination of fluticasone propionate and salmeterol in doses (100 + 50) mcg, (250 + 50) mcg, (500 + 50) mcg administered via the Elpenhaler®
* Patients who should be diagnosed with severe COPD and FEV1 <60% of the expected normal rate and a history of repeated exacerbations that have significant symptoms despite regular bronchodilator therapy:

  1. Single LABA bronchoconstriction
  2. Under dual bronchoconstriction LABA / LAMA
  3. Never have received inhaled or systemic corticosteroids (ICS)
  4. Previous ICS use in the past may be present, as long as the patient is not in the same treatment for the last three months.
* Male or female patients over 18 years of age
* Compliance with treatment
* Compliance with study procedures
* Signed informed consent form

Exclusion Criteria:

* Men or women under 18 years of age
* Non-compliance with treatment
* Inappropriate use of inhaled therapies
* Non-compliance in study procedures
* Unsigned patient consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Compliance | 3 months
  Change in MMAS-8 item scale

SECONDARY OUTCOMES:
Quality of Life | 3 months
  Change in CCQ scale

CONTACTS AND LOCATIONS:
Locations (1):
- Evagelismos hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided